CLINICAL TRIAL: NCT03792672
Title: A Randomized, Double-blind, Placebo-Controlled, 3-Period Crossover Study Followed by 1 Open-label Comparator Period to Evaluate Central Nervous System Pharmacodynamic Activity of TAK-653 in Healthy Volunteers Using Transcranial Magnetic Stimulation
Brief Title: A Study to Evaluate Central Nervous System (CNS) Pharmacodynamic Activity of TAK-653 in Healthy Participants Using Transcranial Magnetic Stimulation (TMS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: TAK-653-1003; U1111-1224-5430 (Other: WHO); 2018-004206-26 (EudraCT Number); NL68394.056.18 (Registry Identifier: CCMO)
Record Dates: First submitted 2019-01-02; First posted 2019-01-03 (Actual); Results first posted 2020-07-02 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: The study is a randomized, crossover 6 sequence study in Treatment Periods 1, 2, and 3.
Who Masked: Participant, Investigator
Masking Description: The study is double blind in Treatment Periods 1, 2, and 3 and open-label in Treatment Period 4.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- TAK-653 6 mg + TAK-653 0.5 mg + Placebo + Ketamine 0.5 mg/kg (Experimental): TAK-653 6 milligram (mg) high dose tablets, orally, once on Day 1 of Treatment Period 1, followed by TAK-653 0.5 mg low dose tablets, orally, once on Day 1 of Treatment Period 2, further followed by TAK-653 placebo-matching tablets, orally, once on Day 1 of Treatment Period 3, followed by Ketamine 0.5 milligram per kilogram (mg/kg), intravenous infusion, once on Day 1 of Treatment Period 4. A washout of 10 to 15 days will be maintained between each treatment period.
  Interventions: Drug: TAK-653; Drug: Placebo; Drug: Ketamine
- TAK-653 6 mg + Placebo + TAK-653 0.5 mg + Ketamine 0.5 mg/kg (Experimental): TAK-653 6 mg high dose tablets, orally, once on Day 1 of Treatment Period 1, followed by TAK-653 placebo-matching tablets, orally, once on Day 1 of Treatment Period 2, further followed by TAK-653 0.5 mg low dose tablets, orally, once on Day 1 of Treatment Period 3, followed by Ketamine 0.5 mg/kg, intravenous infusion, once on Day 1 of Treatment Period 4. A washout of 10 to 15 days will be maintained between each treatment period.
  Interventions: Drug: TAK-653; Drug: Placebo; Drug: Ketamine
- TAK-653 0.5 mg + TAK-653 6 mg + Placebo + Ketamine 0.5 mg/kg (Experimental): TAK-653 0.5 mg low dose tablets, orally, once on Day 1 of Treatment Period 1, followed by TAK-653 6 mg high dose tablets, orally, once on Day 1 of Treatment Period 2, further followed by TAK-653 placebo-matching tablets, orally, once on Day 1 of Treatment Period 3, followed by Ketamine 0.5 mg/kg, intravenous infusion, once on Day 1 of Treatment Period 4. A washout of 10 to 15 days will be maintained between each treatment period.
  Interventions: Drug: TAK-653; Drug: Placebo; Drug: Ketamine
- TAK-653 0.5 mg + Placebo + TAK-653 6 mg + Ketamine 0.5 mg/kg (Experimental): TAK-653 0.5 mg low dose tablets, orally, once on Day 1 of Treatment Period 1, followed by TAK-653 placebo-matching tablets, orally, once on Day 1 of Treatment Period 2, further followed by TAK-653 6 mg high dose tablets, orally, once on Day 1 of Treatment Period 3, followed by Ketamine 0.5 mg/kg, intravenous infusion, once on Day 1 of Treatment Period 4. A washout of 10 to 15 days will be maintained between each treatment period.
  Interventions: Drug: TAK-653; Drug: Placebo; Drug: Ketamine
- Placebo + TAK-653 0.5 mg + TAK-653 6 mg + Ketamine 0.5 mg/kg (Experimental): TAK-653 placebo-matching tablets, orally, once on Day 1 of Treatment Period 1, followed by TAK-653 0.5 mg low dose tablets, orally, once on Day 1 of Treatment Period 2, further followed by TAK-653 6 mg high dose tablets, orally, once on Day 1 of Treatment Period 3, followed by Ketamine 0.5 mg/kg, intravenous infusion, once on Day 1 of Treatment Period 4. A washout of 10 to 15 days will be maintained between each treatment period.
  Interventions: Drug: TAK-653; Drug: Placebo; Drug: Ketamine
- Placebo + TAK-653 6 mg + TAK-653 0.5 mg + Ketamine 0.5 mg/kg (Experimental): TAK-653 placebo-matching tablets, orally, once on Day 1 of Treatment Period 1, followed by TAK-653 6 mg high dose tablets, orally, once on Day 1 of Treatment Period 2, further followed by TAK-653 0.5 mg low dose tablets, orally, once on Day 1 of Treatment Period 3, followed by Ketamine 0.5 mg/kg, intravenous infusion, once on Day 1 of Treatment Period 4. A washout of 10 to 15 days will be maintained between each treatment period.
  Interventions: Drug: TAK-653; Drug: Placebo; Drug: Ketamine

INTERVENTIONS:
Drug: TAK-653 — TAK-653 tablets.
Drug: Placebo — TAK-653 placebo-matching tablets.
Drug: Ketamine — Ketamine intravenous infusion.

SUMMARY:
The primary purpose of this study is to determine whether TAK-653, in comparison to placebo, increases CNS excitability, assessed with TMS-evoked motor-evoked potential (MEP) in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-653. This study is designed to evaluate the central pharmacodynamic activity of TAK-653 using TMS. The study will enroll approximately 24 participants to yield 22 participants that complete treatment periods 1, 2, and 3. Participants will be randomly assigned to 1 of the 6 sequences to receive TAK-653 0.5 mg low dose or TAK-653 6 mg high dose or Placebo in double-blind treatment periods 1, 2, and 3, followed by Ketamine 0.5 mg/kg in open-label Treatment period 4.

All participants will receive one dose of TAK-653 (0.5 or 6 mg), or Placebo or Ketamine on Day 1 of each treatment period.

This single center trial will be conducted in the Netherlands. The overall time to participate in this study is 15 weeks. Participants will make 5 visits to the clinic. A washout period of minimum 10 days will be maintained between the doses in treatment periods 1 to 3. Follow-up phone call will be made on Day 14.

ELIGIBILITY:
Inclusion Criteria:

1. Must be judged to be in good health by the investigator, based on clinical evaluations including laboratory safety tests, medical history, physical examination, 12-lead electrocardiogram (ECG), and vital sign measurements performed at the screening visit and before the first dose of study drug.
2. Must be male or female (of nonchildbearing potential) aged 18 to 55 years, inclusive, at the screening visit.
3. Must have a body mass index (BMI) greater than or equal to (>=) 18.5 and less than or equal to (<=) 30.0 kilogram per square meter (kg/m^2) at the screening visit.

Exclusion Criteria:

1. Has a positive alcohol or drug screen.
2. Had major surgery or donated or lost 1 unit of blood (approximately 500 milliliter [mL]) within 4 weeks before the screening visit.
3. Has a history of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to the following: beer [354 mL/12 ounce (oz)], wine [118 mL/4 oz], or distilled spirits [29.5 mL/1 oz] per day).
4. Who regularly smoke more than 5 cigarettes daily or equivalent and unable or unwilling not to smoke during the in-house period.
5. Consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
6. Has a previous or current clinically significant psychiatric disorder according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, (DSM-5) including substance use disorder.
7. Has a history of intracranial mass lesion, hydrocephalus and/or head injury or trauma.
8. Has metal objects in brain or skull.
9. Has a cochlear implant or deep brain stimulation device.
10. Has a history of epilepsy, seizures, or convulsions.
11. Has a family history of epilepsy, seizures, or convulsions.
12. Has abnormal sleeping patterns (example, working night shifts)
13. Has an rMT of more than 75% of the maximum stimulator output, measured using TMS-electromyogram (EMG) during screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- CHDR, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Dijkstra F, O'Donnell P, Klaassen E, Buhl D, Asgharnejad M, Rosen L, Zuiker R, van Gerven J, Jacobs G. Central nervous system effects of TAK-653, an investigational alpha-amino-3-hydroxy-5-methyl-4-isoxazole receptor (AMPAR) positive allosteric modulator in healthy volunteers. Transl Psychiatry. 2022 Sep 24;12(1):408. doi: 10.1038/s41398-022-02148-w. PMID 36153330

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Netherlands from 11 February 2019 to 18 June 2019.
Pre-assignment Details: Healthy participants were enrolled in 1 of the 6 treatment sequences of this 3-period crossover study to receive TAK 653 0.5 milligram (mg) (Low dose), TAK-653 6 mg (high dose), placebo in Treatment Periods 1 to 3, and ketamine 0.5 milligram per kilogram (mg/kg) in an open label treatment Period 4.
Groups:
- Placebo + TAK-653 0.5 mg + TAK-653 6 mg + Ketamine 0.5 mg/kg: TAK-653 placebo-matching tablets, orally, once on Day 1 of Treatment Period 1, followed by TAK-653 0.5 mg low dose tablets, orally, once on Day 1 of Treatment Period 2, further followed by TAK-653 6 mg high dose tablets, orally, once on Day 1 of Treatment Period 3, followed by Ketamine 0.5 mg/kg, infusion, intravenously, once on Day 1 of Treatment Period 4. A Washout Period of at least 10 days was maintained between each treatment period.
- Placebo + TAK-653 6 mg + TAK-653 0.5 mg + Ketamine 0.5 mg/kg: TAK-653 placebo-matching tablets, orally, once on Day 1 of Treatment Period 1, followed by TAK-653 6 mg high dose tablets, orally, once on Day 1 of Treatment Period 2, further followed by TAK-653 0.5 mg low dose tablets, orally, once on Day 1 of Treatment Period 3, followed by Ketamine 0.5 mg/kg, infusion, intravenously, once on Day 1 of Treatment Period 4. A Washout Period of at least 10 days was maintained between each treatment period.
- TAK-653 0.5 mg + Placebo + TAK-653 6 mg + Ketamine 0.5 mg/kg: TAK-653 0.5 mg low dose tablets, orally, once on Day 1 of Treatment Period 1, followed by TAK-653 placebo-matching tablets, orally, once on Day 1 of Treatment Period 2, further followed by TAK-653 6 mg high dose tablets, orally, once on Day 1 of Treatment Period 3, followed by Ketamine 0.5 mg/kg, infusion, intravenously, once on Day 1 of Treatment Period 4. A Washout Period of at least 10 days was maintained between each treatment period.
- TAK-653 0.5 mg + TAK-653 6 mg + Placebo + Ketamine 0.5 mg/kg: TAK-653 0.5 mg low dose tablets, orally, once on Day 1 of Treatment Period 1, followed by TAK-653 6 mg high dose tablets, orally, once on Day 1 of Treatment Period 2, further followed by TAK-653 placebo-matching tablets, orally, once on Day 1 of Treatment Period 3, followed by Ketamine 0.5 mg/kg, infusion, intravenously, once on Day 1 of Treatment Period 4. A Washout Period of at least 10 days was maintained between each treatment period.
- TAK-653 6 mg + Placebo + TAK-653 0.5 mg + Ketamine 0.5 mg/kg: TAK-653 6 mg high dose tablets, orally, once on Day 1 of Treatment Period 1, followed by TAK-653 placebo-matching tablets, orally, once on Day 1 of Treatment Period 2, further followed by TAK-653 0.5 mg low dose tablets, orally, once on Day 1 of Treatment Period 3, followed by Ketamine 0.5 mg/kg, infusion, intravenously, once on Day 1 of Treatment Period 4. A Washout Period of at least 10 days was maintained between each treatment period.
- TAK-653 6 mg + TAK-653 0.5 mg + Placebo + Ketamine 0.5 mg/kg: TAK-653 6 mg high dose tablets, orally, once on Day 1 of Treatment Period 1, followed by TAK-653 0.5 mg low dose tablets, orally, once on Day 1 of Treatment Period 2, further followed by TAK-653 placebo-matching tablets, orally, once on Day 1 of Treatment Period 3, followed by Ketamine 0.5 mg/kg, infusion, intravenously, once on Day 1 of Treatment Period 4. A Washout Period of at least 10 days was maintained between each treatment period.
Period: Treatment Period 1 (1 Day)
Arm/Group | Placebo + TAK-653 0.5 mg + TAK-653 6 mg + Ketamine 0.5 mg/kg | Placebo + TAK-653 6 mg + TAK-653 0.5 mg + Ketamine 0.5 mg/kg | TAK-653 0.5 mg + Placebo + TAK-653 6 mg + Ketamine 0.5 mg/kg | TAK-653 0.5 mg + TAK-653 6 mg + Placebo + Ketamine 0.5 mg/kg | TAK-653 6 mg + Placebo + TAK-653 0.5 mg + Ketamine 0.5 mg/kg | TAK-653 6 mg + TAK-653 0.5 mg + Placebo + Ketamine 0.5 mg/kg
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1 (10 Days)
Arm/Group | Placebo + TAK-653 0.5 mg + TAK-653 6 mg + Ketamine 0.5 mg/kg | Placebo + TAK-653 6 mg + TAK-653 0.5 mg + Ketamine 0.5 mg/kg | TAK-653 0.5 mg + Placebo + TAK-653 6 mg + Ketamine 0.5 mg/kg | TAK-653 0.5 mg + TAK-653 6 mg + Placebo + Ketamine 0.5 mg/kg | TAK-653 6 mg + Placebo + TAK-653 0.5 mg + Ketamine 0.5 mg/kg | TAK-653 6 mg + TAK-653 0.5 mg + Placebo + Ketamine 0.5 mg/kg
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (1 Day)
Arm/Group | Placebo + TAK-653 0.5 mg + TAK-653 6 mg + Ketamine 0.5 mg/kg | Placebo + TAK-653 6 mg + TAK-653 0.5 mg + Ketamine 0.5 mg/kg | TAK-653 0.5 mg + Placebo + TAK-653 6 mg + Ketamine 0.5 mg/kg | TAK-653 0.5 mg + TAK-653 6 mg + Placebo + Ketamine 0.5 mg/kg | TAK-653 6 mg + Placebo + TAK-653 0.5 mg + Ketamine 0.5 mg/kg | TAK-653 6 mg + TAK-653 0.5 mg + Placebo + Ketamine 0.5 mg/kg
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (10 Days)
Arm/Group | Placebo + TAK-653 0.5 mg + TAK-653 6 mg + Ketamine 0.5 mg/kg | Placebo + TAK-653 6 mg + TAK-653 0.5 mg + Ketamine 0.5 mg/kg | TAK-653 0.5 mg + Placebo + TAK-653 6 mg + Ketamine 0.5 mg/kg | TAK-653 0.5 mg + TAK-653 6 mg + Placebo + Ketamine 0.5 mg/kg | TAK-653 6 mg + Placebo + TAK-653 0.5 mg + Ketamine 0.5 mg/kg | TAK-653 6 mg + TAK-653 0.5 mg + Placebo + Ketamine 0.5 mg/kg
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (1 Day)
Arm/Group | Placebo + TAK-653 0.5 mg + TAK-653 6 mg + Ketamine 0.5 mg/kg | Placebo + TAK-653 6 mg + TAK-653 0.5 mg + Ketamine 0.5 mg/kg | TAK-653 0.5 mg + Placebo + TAK-653 6 mg + Ketamine 0.5 mg/kg | TAK-653 0.5 mg + TAK-653 6 mg + Placebo + Ketamine 0.5 mg/kg | TAK-653 6 mg + Placebo + TAK-653 0.5 mg + Ketamine 0.5 mg/kg | TAK-653 6 mg + TAK-653 0.5 mg + Placebo + Ketamine 0.5 mg/kg
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3 (10 Days)
Arm/Group | Placebo + TAK-653 0.5 mg + TAK-653 6 mg + Ketamine 0.5 mg/kg | Placebo + TAK-653 6 mg + TAK-653 0.5 mg + Ketamine 0.5 mg/kg | TAK-653 0.5 mg + Placebo + TAK-653 6 mg + Ketamine 0.5 mg/kg | TAK-653 0.5 mg + TAK-653 6 mg + Placebo + Ketamine 0.5 mg/kg | TAK-653 6 mg + Placebo + TAK-653 0.5 mg + Ketamine 0.5 mg/kg | TAK-653 6 mg + TAK-653 0.5 mg + Placebo + Ketamine 0.5 mg/kg
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 3 | 4 | 3 | 2 | 4 | 4
Not Completed | 1 | 0 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Period: Treatment Period 4 (2 Days)
Arm/Group | Placebo + TAK-653 0.5 mg + TAK-653 6 mg + Ketamine 0.5 mg/kg | Placebo + TAK-653 6 mg + TAK-653 0.5 mg + Ketamine 0.5 mg/kg | TAK-653 0.5 mg + Placebo + TAK-653 6 mg + Ketamine 0.5 mg/kg | TAK-653 0.5 mg + TAK-653 6 mg + Placebo + Ketamine 0.5 mg/kg | TAK-653 6 mg + Placebo + TAK-653 0.5 mg + Ketamine 0.5 mg/kg | TAK-653 6 mg + TAK-653 0.5 mg + Placebo + Ketamine 0.5 mg/kg
Started | 3 | 4 | 3 | 2 | 4 | 4
Completed | 2 | 4 | 3 | 2 | 4 | 4
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug. Baseline characteristics data has been presented for overall participants analyzed.
Groups:
- All Participants: TAK-653 placebo-matching tablets or TAK-653 0.5 mg low dose tablets or TAK-653 6 mg high dose tablets, orally, once, on Day 1 of respective Treatment Period 1, 2 or 3 and Ketamine 0.5 mg/kg, infusion, intravenously, once on Day 1 of Treatment Period 4. A Washout Period of at least 10 days was maintained between each treatment period.
Arm/Group | All Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 24
Weight [Mean (Standard Deviation); unit: kilogram (Kg)] | 79.12 (10.81)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 181.98 (9.88)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 23.93 (2.85)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Peak-to-Peak Amplitude of Motor-evoked Potential (MEP) Obtained With Single-pulse Transcranial Magnetic Stimulation (TMS) for TAK-653 at 2.5 Hours Post TAK-653 Dose
Description: TMS was a neurophysiologic test for assessing upper motor neuron function. TMS was a noninvasive neuro stimulation method involving the application of brief magnetic pulses to the skull, based on the principles of electromagnetic induction, create an orthogonal electric current that can be sufficient to depolarize neurons and activate neuronal circuits. Single-pulse TMS was used to determine peak-to-peak amplitude of MEP at a stimulation intensity of 120 percent (%) of baseline resting motor threshold (rMT). rMT was defined as the minimum stimulus intensity to evoke an MEP. Change in peak-to peak amplitude of MEP was be assessed by TMS after treatment with 0.5 mg or 6 mg of TAK-653 versus (vs.) matched oral placebo.
Time Frame: Baseline, 2.5 hours post TAK-653 dose
Population: The pharmacodynamics (PD) set included of all participants who received study drug and had at least one postdose PD measurement. The PD analysis set included all participants who had completed first 3 treatment periods. Participants who were evaluable for this measure at given time point were included for the assessment.
Measure: Mean (Standard Deviation); unit: microvolt (mcV)
Groups:
- Placebo: TAK-653 placebo-matching tablets, orally, once on Day 1 of Treatment Period 1, 2 or 3 as per assigned treatment sequence.
- TAK-653 0.5 mg: TAK-653 0.5 mg low dose tablets, orally, once on Day 1 of Treatment Period 1, 2 or 3 as per assigned treatment sequence.
- TAK-653 6 mg: TAK-653 6 mg high dose tablets, orally, once on Day 1 of Treatment Period 1, 2 or 3 as per assigned treatment sequence.
Arm/Group | Placebo | TAK-653 0.5 mg | TAK-653 6 mg
Number analyzed (Participants) | 24 | 24 | 24
microvolt (mcV)
  Baseline: number analyzed (Participants) | 24 | 24 | 23
  Baseline | 898.828 (693.1535) | 841.068 (591.1367) | 1004.127 (574.5982)
  Change at 2.5 Hours Post TAK-653 Dose: number analyzed (Participants) | 24 | 24 | 23
  Change at 2.5 Hours Post TAK-653 Dose | -139.117 (829.5901) | 17.265 (466.2556) | 139.932 (813.9705)
Statistical Analysis 1: Comparison: Placebo vs TAK-653 0.5 mg; Test type: Superiority; p = 0.4278, Mixed Models Analysis — Based on mixed model analysis, with treatment, period, sequence, treatment-by-period interaction as fixed factors, participant within sequence as a random factor, baseline as a covariate; Least square mean (LSM) difference = 115, 90% CI 2-sided [-128 to 359], Standard Error of Mean 144
Statistical Analysis 2: Comparison: Placebo vs TAK-653 6 mg; Test type: Superiority; p = 0.0269, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LSM difference = 338, 90% CI 2-sided [90.5 to 585], Standard Error of Mean 147

2. Primary Outcome: Change From Baseline in Resting Motor Threshold (rMT) Obtained With Single-pulse TMS for TAK-653 at 2.5 Hours Post TAK-653 Dose
Description: The rMT was defined as the minimum stimulus intensity to evoke an MEP. Single-pulse TMS was used to determine rMT. A lower rMT value indicated greater neuronal excitability. TMS was a neurophysiologic test for assessing upper motor neuron function. TMS was a noninvasive neuro stimulation method involving the application of brief magnetic pulses to the skull, based on the principles of electromagnetic induction, create an orthogonal electric current that can be sufficient to depolarize neurons and activate neuronal circuits. Change in rMT was be assessed by TMS after treatment with 0.5 mg or 6 mg of TAK-653 vs. matched oral placebo.
Time Frame: Baseline, 2.5 hours post TAK-653 dose
Population: The PD set included of all participants who received study drug and had at least one postdose PD measurement. The PD analysis set included all participants who had completed first 3 treatment periods.
Measure: Mean (Standard Deviation); unit: percentage of maximum stimulator output
Arm/Group | Placebo | TAK-653 0.5 mg | TAK-653 6 mg
Number analyzed (Participants) | 24 | 24 | 24
percentage of maximum stimulator output
  Baseline | 55.3 (7.46) | 55.9 (8.99) | 55.3 (8.93)
  Change at 2.5 hours post TAK-653 Dose | -0.1 (2.74) | -0.5 (1.74) | -0.3 (1.95)
Statistical Analysis 1: Comparison: Placebo vs TAK-653 0.5 mg; Test type: Superiority; p = 0.5089, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LSM difference = -0.388, 90% CI 2-sided [-1.37 to 0.595], Standard Error of Mean 0.582
Statistical Analysis 2: Comparison: Placebo vs TAK-653 6 mg; Test type: Superiority; p = 0.7208, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LSM difference = -0.209, 90% CI 2-sided [-1.19 to 0.773], Standard Error of Mean 0.581

3. Secondary Outcome: Change From Baseline in Magnitude of Long Intracortical Inhibition (LICI) Obtained With Paired-pulse TMS for TAK-653 at 2.5 Hours Post TAK-653 Dose
Description: LICI was TMS stimulation paradigm that capture modulation of cortical excitation-inhibition balance with pairs of TMS pulses at stimulation intensity conditioning pulse and test pulse of 120% of baseline rMT. rMT was defined as the minimum stimulus intensity to evoke an MEP. TMS was a neurophysiologic test for assessing upper motor neuron function. TMS was a noninvasive neuro stimulation method involving the application of brief magnetic pulses to the skull, based on the principles of electromagnetic induction, create an orthogonal electric current that can be sufficient to depolarize neurons and activate neuronal circuits. Change in LICI was be assessed by TMS after treatment with 0.5 mg or 6 mg of TAK-653 vs. matched oral placebo.
Time Frame: Baseline, 2.5 hours post TAK-653 dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent inhibition
Arm/Group | Placebo | TAK-653 0.5 mg | TAK-653 6 mg
Number analyzed (Participants) | 24 | 24 | 24
percent inhibition
  Baseline: LICI 50 ms | 75.113 (97.2865) | 96.515 (113.2728) | 96.568 (111.1657)
  Change at 2.5 Hours Post TAK-653 Dose: LICI 50 ms | 0.675 (54.5725) | 18.319 (81.4378) | 19.395 (110.0870)
  Baseline: LICI 100 ms | 16.167 (27.0976) | 10.430 (14.1289) | 46.808 (149.9806)
  Change at 2.5 Hours Post TAK-653 Dose: LICI 100 ms | 0.147 (29.1567) | 5.905 (18.8939) | -28.644 (142.5618)
  Baseline: LICI 200 ms | 48.149 (33.1815) | 48.934 (48.6073) | 49.773 (37.7173)
  Change at 2.5 Hours Post TAK-653 Dose: LICI 200 ms | 2.882 (21.2459) | 9.902 (42.5761) | 11.540 (30.1594)
  Baseline: LICI 300 ms | 59.463 (31.1596) | 56.115 (36.8452) | 54.572 (30.5543)
  Change at 2.5 Hours Post TAK-653 Dose: LICI 300 ms | -9.996 (27.7151) | 8.618 (36.0453) | 1.638 (32.6843)
Statistical Analysis 1: Comparison: Placebo vs TAK-653 0.5 mg; LICI 50 ms peak-to-peak amplitude; Test type: Superiority; p = 0.4174, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LSM difference = 14.0, 90% CI 2-sided [-14.8 to 42.8], Standard Error of Mean 17.1
Statistical Analysis 2: Comparison: Placebo vs TAK-653 6 mg; LICI 50 ms peak-to-peak amplitude; Test type: Superiority; p = 0.3832, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LSM difference = 15.1, 90% CI 2-sided [-25.3 to 31.5], Standard Error of Mean 17.1
Statistical Analysis 3: Comparison: Placebo vs TAK-653 0.5 mg; LICI 100 ms peak-to-peak amplitude; Test type: Superiority; p = 0.9368, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LSM difference = -0.326, 90% CI 2-sided [-7.23 to 6.58], Standard Error of Mean 4.09
Statistical Analysis 4: Comparison: Placebo vs TAK-653 6 mg; LICI 100 ms peak-to-peak amplitude; Test type: Superiority; p = 0.3790, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LSM difference = 3.71, 90% CI 2-sided [-3.32 to 10.7], Standard Error of Mean 4.16
Statistical Analysis 5: Comparison: Placebo vs TAK-653 0.5 mg; LICI 200 ms peak-to-peak amplitude; Test type: Superiority; p = 0.2580, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LSM difference = 7.36, 90% CI 2-sided [-3.44 to 18.2], Standard Error of Mean 6.41
Statistical Analysis 6: Comparison: Placebo vs TAK-653 6 mg; LICI 200 ms peak-to-peak amplitude; Test type: Superiority; p = 0.1524, Mixed Models Analysis; LSM difference = 9.36, 90% CI 2-sided [-1.45 to 20.2], Standard Error of Mean 6.41
Statistical Analysis 7: Comparison: Placebo vs TAK-653 0.5 mg; LICI 300 ms peak-to-peak amplitude; Test type: Superiority; p = 0.0220, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LSM difference = 17.2, 90% CI 2-sided [5.06 to 29.4], Standard Error of Mean 7.21
Statistical Analysis 8: Comparison: Placebo vs TAK-653 6 mg; LICI 300 ms peak-to-peak amplitude; Test type: Superiority; p = 0.1927, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LSM difference = 9.58, 90% CI 2-sided [-2.59 to 21.8], Standard Error of Mean 7.23

4. Secondary Outcome: Change From Baseline in Magnitude of Short Intracortical Inhibition (SICI) Obtained With Paired-pulse TMS for TAK-653 at 2.5 Hours Post TAK-653 Dose
Description: SICI was TMS stimulation paradigm that capture modulation of cortical excitation-inhibition balance with pairs of TMS pulses at stimulation intensity conditioning pulse 80% of baseline rMT and test pulse of 120% of baseline rMT. rMT was defined as the minimum stimulus intensity to evoke an MEP. TMS was a neurophysiologic test for assessing upper motor neuron function. TMS was a noninvasive neuro stimulation method involving the application of brief magnetic pulses to the skull, based on the principles of electromagnetic induction, create an orthogonal electric current that can be sufficient to depolarize neurons and activate neuronal circuits. Change in SICI was be assessed by TMS after treatment with 0.5 mg or 6 mg of TAK-653 vs. matched oral placebo.
Time Frame: Baseline, 2.5 hours post TAK-653 dose
Population: The PD set included of all participants who received study drug and had at least one postdose PD measurement. The PD analysis set included all participants who had completed first 3 treatment periods. Participants who were evaluable for this measure at given time point were included for the assessment.
Measure: Mean (Standard Deviation); unit: percent inhibition
Arm/Group | Placebo | TAK-653 0.5 mg | TAK-653 6 mg
Number analyzed (Participants) | 24 | 24 | 24
percent inhibition
  Baseline: SICI 2 ms: number analyzed (Participants) | 24 | 24 | 23
  Baseline: SICI 2 ms | 43.095 (30.7011) | 39.159 (39.2536) | 47.951 (42.1139)
  Change at 2.5 Hours Post TAK-653 Dose: SICI 2 ms: number analyzed (Participants) | 24 | 24 | 23
  Change at 2.5 Hours Post TAK-653 Dose: SICI 2 ms | 5.052 (47.5676) | 1.772 (35.9158) | -14.580 (37.7311)
  Baseline: SICI 5 ms: number analyzed (Participants) | 24 | 24 | 23
  Baseline: SICI 5 ms | 70.640 (49.8699) | 59.672 (37.7419) | 72.722 (62.0484)
  Change at 2.5 Hours Post TAK-653 Dose: SICI 5 ms | 14.303 (81.6111) | 4.274 (30.8966) | -7.247 (52.9205)
Statistical Analysis 1: Comparison: Placebo vs TAK-653 0.5 mg; SICI 2 ms peak-to-peak amplitude; Test type: Superiority; p = 0.5590, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LSM difference = -5.65, 90% CI 2-sided [-21.8 to 10.5], Standard Error of Mean 9.59
Statistical Analysis 2: Comparison: Placebo vs TAK-653 6 mg; SICI 2 ms peak-to-peak amplitude; Test type: Superiority; p = 0.1049, Mixed Models Analysis; LSM difference = -16.1, 90% CI 2-sided [-32.5 to 0.242], Standard Error of Mean 9.72
Statistical Analysis 3: Comparison: Placebo vs TAK-653 0.5 mg; SICI 5 ms peak-to-peak amplitude; Test type: Superiority; p = 0.2238, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LSM difference = -16.7, 90% CI 2-sided [-39.4 to 6.06], Standard Error of Mean 13.5
Statistical Analysis 4: Comparison: Placebo vs TAK-653 6 mg; SICI 5 ms peak-to-peak amplitude; Test type: Superiority; p = 0.1847, Mixed Models Analysis; LSM difference = -18.3, 90% CI 2-sided [-41.3 to 4.56], Standard Error of Mean 13.6

5. Secondary Outcome: Change From Baseline in rMT Obtained With Single-pulse TMS to Assess the Effect of Ketamine at 2.5 Hours and 24 Hours Post-dose of Ketamine
Description: The rMT was defined as the minimum stimulus intensity to evoke an MEP. Single-pulse TMS was used to determine rMT. A lower rMT value indicated greater neuronal excitability. TMS was a neurophysiologic test for assessing upper motor neuron function. TMS was a noninvasive neuro stimulation method involving the application of brief magnetic pulses to the skull, based on the principles of electromagnetic induction, create an orthogonal electric current that can be sufficient to depolarize neurons and activate neuronal circuits. Change in rMT was be assessed by TMS after treatment with 0.5 mg/kg Ketamine.
Time Frame: Baseline, 2.5 hours post ketamine dose, and 24 hours post ketamine dose
Population: The PD set included of all participants who received study drug and had at least one postdose PD measurement. The PD analysis set included all participants who had completed Treatment Period 4. Participants who were evaluable for this measure at given time point were included for the assessment.
Measure: Mean (Standard Deviation); unit: percentage of maximum stimulator output
Groups:
- Ketamine 0.5 mg/kg: Ketamine 0.5 mg/kg, infusion, intravenously, once on Day 1 of Treatment Period 4 in all 6 treatment sequences.
Arm/Group | Ketamine 0.5 mg/kg
Number analyzed (Participants) | 20
percentage of maximum stimulator output
  Baseline | 54.4 (9.28)
  Change at 2.5 hours Ketamine Post Dose: number analyzed (Participants) | 19
  Change at 2.5 hours Ketamine Post Dose | 0.7 (4.18)
  Change at 24 hours Ketamine Post Dose: number analyzed (Participants) | 19
  Change at 24 hours Ketamine Post Dose | 0.8 (3.10)

6. Secondary Outcome: Change From Baseline in in Peak-to-Peak Amplitude of MEP Obtained With Single-pulse TMS to Assess the Effect of Ketamine at 2.5 Hours and 24 Hours Post Dose of Ketamine
Description: TMS was a neurophysiologic test for assessing upper motor neuron function. TMS was a noninvasive neuro stimulation method involving the application of brief magnetic pulses to the skull, based on the principles of electromagnetic induction, create an orthogonal electric current that can be sufficient to depolarize neurons and activate neuronal circuits. Single-pulse TMS was used to determine peak-to-peak amplitude of MEP at a stimulation intensity of 120% of baseline rMT. rMT was defined as the minimum stimulus intensity to evoke an MEP. Change in peak-to peak amplitude of MEP was be assessed by TMS after treatment 0.5 mg/kg Ketamine.
Time Frame: Baseline, 2.5 hours post ketamine dose, and 24 hours post ketamine dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mcV
Arm/Group | Ketamine 0.5 mg/kg
Number analyzed (Participants) | 20
mcV
  Baseline | 1150.618 (1047.3920)
  Change at 2.5 hours Ketamine Post Dose: number analyzed (Participants) | 19
  Change at 2.5 hours Ketamine Post Dose | -193.897 (897.0245)
  Change at 24 hours Ketamine Post Dose: number analyzed (Participants) | 18
  Change at 24 hours Ketamine Post Dose | -295.041 (944.4889)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug until 14 days after last dose in Treatment Period 4 (up to Day 48)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | TAK-653 0.5 mg | TAK-653 6 mg | Ketamine 0.5 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/20
Other Adverse Events (participants affected / at risk) | 7/24 | 9/24 | 12/24 | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | TAK-653 0.5 mg (N=24) | TAK-653 6 mg (N=24) | Ketamine 0.5 mg/kg (N=20)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 8 (8)
Headache (Nervous system disorders) | 2 (3) | 1 (1) | 4 (4) | 3 (3)
Somnolence (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3) | 3 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Feeling Cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Feeling Drunk (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Seasonal Allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dissociation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT03792672/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/72/NCT03792672/SAP_001.pdf